CLINICAL TRIAL: NCT01044719
Title: What Duration of Intravenous Antibiotic Therapy Should be Used in the Treatment of Infective Exacerbations of Cystic Fibrosis Chronically Colonised With Pseudomonas Aeruginosa
Brief Title: Duration of Antibiotics in Infective Exacerbations of Cystic Fibrosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Prof Margaret Hodson, Imperial College London
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RBHADS001
Record Dates: First submitted 2009-12-14; First posted 2010-01-08 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ceftazidime; Tobramycin; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 days (Active Comparator)
  Interventions: Drug: Ceftazidime; Drug: Tobramycin; Drug: Meropenem
- 14 days (Active Comparator)
  Interventions: Drug: Ceftazidime; Drug: Tobramycin; Drug: Meropenem
- 21 days (Active Comparator)
  Interventions: Drug: Ceftazidime; Drug: Tobramycin; Drug: Meropenem

INTERVENTIONS:
Drug: Ceftazidime — Ceftazidime 2g TDS IV
Drug: Tobramycin — Tobramycin 7mg/kg/day OD IV
Drug: Meropenem — Meropenem 2g TDS IV

SUMMARY:
Cystic Fibrosis patients attending with infective exacerbations will be enrolled into the study. The trial is a double blinded, randomised trial with patients randomised to 10,14 or 21 days of antibiotic therapy, comprising of tobramycin and either ceftazidime or meropenem.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Diagnosis of Cystic Fibrosis
* Presenting with Infective exacerbation

Exclusion Criteria:

* Unable to give consent
* Allergy to study medications
* Intolerance of aminoglycoside antibiotics
* Pseudomonas resistant to study antibiotics
* On the active transplant list or FEV1<20% predicted
* Pregnancy/breast-feeding
* Co-existent ABPA requiring a change in treatment
* Co-existent mycobacterial infection
* A previous participant in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-10 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Treatment failure at completion of antibiotic course | 21 days
Time to next exacerbation | 6 months

SECONDARY OUTCOMES:
Change in Spirometry | up to 21 days
Change in inflammatory markers | up to 21 days
Change in sputum bacteriology | up to 21 days
Adverse effects of study antibiotics | Up to 21 days
Quality of life scores | Up to 21 days
Change in nutritional status | up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hodson, MD FRCP DA, Principal Investigator — Imperial College London
Locations (1):
- Department of Cystic Fibrosis, Royal Brompton Hospital, London, United Kingdom